CLINICAL TRIAL: NCT01224782
Title: Evaluation of Treatment With Zemplar Capsules in the Therapy of Secondary Hyperparathyroidism (SHPT) in Subjects With Chronic Kidney Disease (CKD) Stage 3 or 4 in the Conditions of Routine Clinical Practice. A Multi-country, Multi-center Post Marketing Observational Study in Routine Clinical Use in Eastern European Countries.
Brief Title: Evaluation of Treatment With Zemplar Capsules in the Therapy of Secondary Hyperparathyroidism (SHPT)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-269
Record Dates: First submitted 2010-09-27; First posted 2010-10-20 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism
Keywords: Zemplar capsules; Chronic kidney disease (CKD) stage 3 or 4; Secondary hyperparathyroidism (SHPT); Postmarketing observational study (PMOS)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease, Secondary Hyperparathyroidism: All eligible participants with chronic kidney disease stage 3 and 4 and secondary hyperparathyroidism treated with Zemplar (paricalcitol) capsules according to the local marketing authorization

SUMMARY:
The aims of this post-marketing observational study (PMOS) are to evaluate the time period needed to achieve > 30% decrease of intact parathyroid hormone (iPTH) compared to the initial values and to provide data on the tolerability and compliance of treatment with Zemplar (paricalcitol) capsules in the therapy of secondary hyperparathyroidism (SHPT) in patients with chronic kidney disease (CKD) stage 3 or 4 in conditions of routine clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional, observational, open-label, multi-country, multicenter post-marketing study in which Zemplar (paricalcitol) is prescribed in the usual manner in accordance with the terms of the local marketing authorization. Follow up visits will occur 1, 3, 6, 9, and 12 months after screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with chronic kidney disease (CKD) stage 3 and 4 and secondary hyperparathyroidism (SHPT)
* Patients with Intact Parathyroid Hormone (iPTH) > 70 pg/mL and with chronic kidney disease (CKD) stage 3 or with Intact Parathyroid Hormone (iPTH) > 110 pg/mL and with chronic kidney disease (CKD) stage 4
* Patients clinically indicated for treatment with Zemplar capsules
* Patient must provide the authorization to use his/her data for statistical evaluation before entering to the post marketing observational study (PMOS). Local Law requirements are to be followed

Exclusion Criteria:

* Patients with clinically important hypercalcemia = Calcium > 2.6 mmol/L (10.5 mg/dL)
* Patients suffering from proved intoxication of vitamin D or patient with known hypersensitivity to paricalcitol or any other part of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Zemplar capsules will be prescribed in usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication as well as local guidelines. The decision to prescribe or not prescribe Zemplar capsules would be made prior to entry of a subject in the study.
  Medical doctors with experience in treatment of patients with chronic kidney disease (CKD) stage 3 or 4 and secondary hyperparathyroidism (SHPT) will observe each enrolled patient for a period of 12 months.
  Follow-up of patients should enable 6 patient visits during this period.
Sampling Method: Non-Probability Sample
Enrollment: 994 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Ionescu, MD, Study Director — AbbVie
Locations (69):
- Bulgaria (9):
  - Site Reference ID/Investigator# 66544, Montana
  - Site Reference ID/Investigator# 47685, Pleven
  - Site Reference ID/Investigator# 66546, Plovdiv
  - Site Reference ID/Investigator# 47683, Sofia
  - Site Reference ID/Investigator# 66543, Sofia
  - Site Reference ID/Investigator# 47684, Sofia
  - Site Reference ID/Investigator# 66542, Sofia
  - Site Reference ID/Investigator# 66545, Sofia
  - Site Reference ID/Investigator# 47687, Varna
- Czechia (28):
  - Site Reference ID/Investigator# 43449, Beroun
  - Site Reference ID/Investigator# 46744, Brno
  - Site Reference ID/Investigator# 73353, Brno
  - Site Reference ID/Investigator# 47690, Brno
  - Site Reference ID/Investigator# 46742, České Budějovice
  - Site Reference ID/Investigator# 49542, Frýdek-Místek
  - Site Reference ID/Investigator# 67442, Jilemnice
  - Site Reference ID/Investigator# 67443, Jilemnice
  - Site Reference ID/Investigator# 51003, Karlovy Vary
  - Site Reference ID/Investigator# 51004, Mariánské Lázně
  - Site Reference ID/Investigator# 43522, Nový Jičín
  - Site Reference ID/Investigator# 43523, Nový Jičín
  - Site Reference ID/Investigator# 43524, Nový Jičín
  - Site Reference ID/Investigator# 45483, Olomouc
  - Site Reference ID/Investigator# 43453, Ostrava
  - Site Reference ID/Investigator# 46743, Pilsen
  - Site Reference ID/Investigator# 51008, Prague
  - Site Reference ID/Investigator# 47842, Prague
  - Site Reference ID/Investigator# 68462, Prague
  - Site Reference ID/Investigator# 51005, Prague
  - Site Reference ID/Investigator# 51009, Prague
  - Site Reference ID/Investigator# 51011, Prague
  - Site Reference ID/Investigator# 48210, Přerov
  - Site Reference ID/Investigator# 45487, Rakovník
  - Site Reference ID/Investigator# 51012, Slaný
  - Site Reference ID/Investigator# 51002, Sokolov
  - Site Reference ID/Investigator# 43448, Trutnov
  - Site Reference ID/Investigator# 45485, Vyškov
- Romania (32):
  - Site Reference ID/Investigator# 42992, Bacau
  - Site Reference ID/Investigator# 42879, Bucharest
  - Site Reference ID/Investigator# 42880, Bucharest
  - Site Reference ID/Investigator# 42881, Bucharest
  - Site Reference ID/Investigator# 42882, Bucharest
  - Site Reference ID/Investigator# 42883, Bucharest
  - Site Reference ID/Investigator# 42963, Bucharest
  - Site Reference ID/Investigator# 42970, Bucharest
  - Site Reference ID/Investigator# 42877, Bucharest
  - Site Reference ID/Investigator# 42878, Bucharest
  - Site Reference ID/Investigator# 42973, Bucharest
  - Site Reference ID/Investigator# 42975, Bucharest
  - Site Reference ID/Investigator# 42976, Bucharest
  - Site Reference ID/Investigator# 42981, Cluj-Napoca
  - Site Reference ID/Investigator# 42982, Cluj-Napoca
  - Site Reference ID/Investigator# 42980, Cluj-Napoca
  - Site Reference ID/Investigator# 63623, Cluj-Napoca
  - Site Reference ID/Investigator# 43009, Constanța
  - Site Reference ID/Investigator# 43002, Craiova
  - Site Reference ID/Investigator# 43003, Craiova
  - Site Reference ID/Investigator# 43006, Craiova
  - Site Reference ID/Investigator# 42991, Iași
  - Site Reference ID/Investigator# 42988, Iași
  - Site Reference ID/Investigator# 42989, Iași
  - Site Reference ID/Investigator# 42999, Oradea
  - Site Reference ID/Investigator# 43000, Oradea
  - Site Reference ID/Investigator# 42979, Ploieşti
  - Site Reference ID/Investigator# 42984, Târgu Mureş
  - Site Reference ID/Investigator# 42985, Târgu Mureş
  - Site Reference ID/Investigator# 42987, Târgu Mureş
  - Site Reference ID/Investigator# 42994, Timișoara
  - Site Reference ID/Investigator# 42995, Timișoara

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Started | 994
Completed | 730
Not Completed | 264
Not completed — Lost to Follow-up | 177
Not completed — Withdrawal by Subject | 16
Not completed — Death | 14
Not completed — Improvement | 13
Not completed — Adverse Event | 12
Not completed — Adverse Reaction | 11
Not completed — Noncompliance | 10
Not completed — Other | 4
Not completed — Start of Dialysis | 3
Not completed — Change of Treatment | 1
Not completed — Financial Reasons | 1
Not completed — Deterioration | 1
Not completed — Transplantation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 994
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.29 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 477
  Male | 517
Baseline Chronic Kidney Disease Stage [Number; unit: percentage of participants] — Stage 3: Glomerular Filtration Rate 30 - 59 mL/min/1.73 m^2; Stage 4: Glomerular Filtration Rate 15 - 29 mL/min/1.73 m^2.
  percentage of participants
    Chronic Kidney Disease Stage 3 | 40.8
    Chronic Kidney Disease Stage 4 | 59.2
Baseline Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pmol/L] | 36.33 (53.7)

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve a > 30% Decrease From Baseline in Intact Parathyroid Hormone (iPTH) Values
Description: Mean time to achieve a > 30% decrease in intact parathyroid hormone (iPTH) compared with the initial values at baseline (screening visit).
Time Frame: From Baseline up to 12 Months
Population: The primary analysis was conducted in the per-protocol (PP) population, which included all participants for whom all study criteria were fulfilled at the time of enrollment and who had no major protocol deviation occur in the course of the study, with a > 30% decrease in iPTH compared with the initial values at baseline.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 694
months | 3.82 (3.37)

2. Primary Outcome: Percentage of Participants With Calcium x Phosphorus Product (CxP) Values > 65 mg˄2/dL˄2 or 5.24 mmol˄2/L˄2
Description: The percentage of participants with Calcium x Phosphorus Product (CxP) values > 65 mg˄2/dL˄2 or 5.24 mmol˄2/L˄2 at any timepoint during followup, up to 12 months.
Time Frame: From Baseline up to 12 Months
Population: The primary analysis was conducted in the per-protocol (PP) population, which included all participants for whom all study criteria were fulfilled at the time of enrollment and who had no major protocol deviation occur in the course of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 919
percentage of participants | 7.4

3. Secondary Outcome: Percentage of Participants Who Achieved a > 30% Decrease From Baseline in Intact Parathyroid Hormone (iPTH)
Description: The percentage of participants with a decrease in iPTH levels > 30% at any timepoint during followup, up to 12 months.
Time Frame: From Baseline up to 12 Months
Population: Secondary analyses were conducted in the intent-to-treat (ITT) population, which included all participants who received at least 1 dose of study drug and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 935
percentage of participants | 75.3

4. Secondary Outcome: Percentage of Participants With Hypercalcemia
Description: The percentage of participants with hypercalcemia (Calcium > 2.6 mmol/L [10.5 mg/dL]) at any timepoint during followup, up to 12 months.
Time Frame: From Baseline up to 12 months
Population: The safety population included all participants who received at least 1 dose of study drug and for whom safety data was collected after administration of the first dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 994
percentage of participants | 0.9

5. Secondary Outcome: Mean Weekly Dose of Zemplar (Paricalcitol)
Description: Compliance was assessed using the mean weekly total dose of Zemplar (paricalcitol).
Time Frame: From Baseline up to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 994
micrograms
  Screening to Month 1 (N=994) | 6.29 (2.49)
  Month 9 to Month 12 (N=737) | 5.77 (3.31)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. An Adverse Drug Reaction (ADR) is any noxious and undesired reaction related to an experimental drug or experiment. A serious adverse event (SAE) is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome. AEs were rated for severity as either Mild: transient and easily tolerated; Moderate: causes discomfort and interrupts usual activities; or Severe: causes considerable interference with usual activities, may be incapacitating or life-threatening. AEs related to Zemplar (paricalcitol) were assessed as being either probably or possibly related by the investigator.
Time Frame: Adverse events were collected from the screening visit to month 12 (total 13 months); Serious Adverse Events were collected from the time that informed consent was obtained to 30 days after last dose of study drug (up to 13 months)
Population: The safety population included all participants who received at least 1 dose of study drug and for whom safety data was collected after administration of the first dose of study drug .
Measure: Number; unit: participants
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Number analyzed (Participants) | 994
participants
  Any AE | 141
  Any Serious AE | 27
  Deaths | 14
  Adverse Events Probably Related | 14
  AEs Possibly Related to Study Drug | 14
  AEs Probably Not Related to Study Drug | 13
  AEs Not Related to Study Drug | 100

ADVERSE EVENTS:
Time Frame: All participants who received at least 1 dose of study drug and for whom safety data was collected after administration of the first dose of study drug.
Arm/Group | Chronic Kidney Disease, Secondary Hyperparathyroidism
Serious Adverse Events (participants affected / at risk) | 27/994
Other Adverse Events (participants affected / at risk) | 66/994
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease, Secondary Hyperparathyroidism (N=994)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 4
Cardiac failure acute (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiorenal syndrome (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Malaise (General disorders) | 1
Pallor (General disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Cardiac amyloidosis (Immune system disorders) | 1
Renal amyloidosis (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Oedema (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Psychiatric symptom (Psychiatric disorders) | 1
Congenital cystic kidney disease (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Haemodialysis (Surgical and medical procedures) | 4
Leg amputation (Surgical and medical procedures) | 1
Renal transplant (Surgical and medical procedures) | 1
Acute myocardial infarction (Vascular disorders) | 3
Atherosclerosis obliterans (Vascular disorders) | 1
Diabetic foot (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive nephropathy (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Myocardial infarction (Vascular disorders) | 2
Pulmonary embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease, Secondary Hyperparathyroidism (N=994)
Nausea (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 5
Pyrexia (General disorders) | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 9
Hyperphosphataemia (Metabolism and nutrition disorders) | 6
Azotaemia (Renal and urinary disorders) | 5
Dysuria (Renal and urinary disorders) | 5
Renal failure chronic (Renal and urinary disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Haemodialysis (Surgical and medical procedures) | 12
Hypertension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.